CLINICAL TRIAL: NCT06542614
Title: A Phase II Clinical Trial to Evaluate the Efficacy, Safety, Pharmacokinetics (PK), and Pharmacodynamic (PD) Profile of TQH3906 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Treatment of Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH3906-II-01
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH3906 capsules (Experimental): TQH3906 capsules are administered orally at the same time (±2 hours) on an empty stomach every day for 12 weeks starting from Day 1.
  Interventions: Drug: TQH3906 capsules
- Placebo of TQH3906 capsules (Placebo Comparator): TQH3906 capsules placebo: TQH3906 capsules placebo administered orally once daily for 12 weeks at the same time (±2 hours) on an empty stomach starting from Day 1.
  Interventions: Drug: Placebo of TQH3906 capsules

INTERVENTIONS:
Drug: TQH3906 capsules — To assess the efficacy and safety of TQH3906 in subjects with moderate to severe plaque psoriasis.
  Arms: TQH3906 capsules
Drug: Placebo of TQH3906 capsules — Placebo without drug substance.
  Arms: Placebo of TQH3906 capsules

SUMMARY:
To assess the efficacy and safety of TQH3906 in subjects with moderate to severe plaque psoriasis, as well as the PK and PD characteristics of multiple doses

ELIGIBILITY:
Inclusion Criteria:

* Be 18-70 years old (both 18 and 70 years old), regardless of gender；
* Clinically diagnosed with stable moderate to severe plaque psoriasis with a history ≥ 6 months (from randomization), and no morphological changes in skin lesions or significant disease outbreaks as assessed by the investigator;
* Appropriate for systemic therapy or phototherapy as judged by the investigator;
* At screening and baseline, the PASI score was ≥ 12 points, the BSA ≥ 10%, and the sPGA ≥ 3 points ;
* Have a full understanding of this study, voluntarily participate in the trial, and have signed a written informed consent form;
* Subjects (including partners) are willing to voluntarily use appropriate and effective contraceptive measures from screening to 3 months after the last dose of study drug.

Exclusion Criteria:

* Pregnant and lactating females;
* Have other forms of psoriasis other than plaque psoriasis (e.g., guttate psoriasis, generalized pustular psoriasis, erythrodermic psoriasis, arthropathic psoriasis);
* Presence of serovirological abnormalities during the screening period:

  1. Active hepatitis, or hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcA positive and Hepatitis B virus (HBV) DNA positive, or Hepatitis C virus (HCV) antibody positive and HCV-RNA positive;
  2. Positive for HIV antibody during the screening period, or have a history of HIV infection in the past;
  3. Positive Treponema pallidum antibody and positive non-Treponema pallidum serum test (RPR or TRUST) during the screening period;
* Have a history of active tuberculosis during the screening period or before, or have latent tuberculosis infection found at screening (refers to T-SPOT positive without clinical manifestations). (Note: Patients with latent tuberculosis infection can be re-screened 1 month after starting prophylaxis according to the guidelines, and in order to continue to participate in the study, patients must agree to continue to complete the prophylactic regimen during the study, but rifampicin treatment should be avoided.) ;
* Has a history of severe herpes zoster or herpes simplex infection, including but not limited to herpetic encephalitis, disseminated herpes simplex, generalized herpes zoster;
* History of severe bacterial, fungal or viral infection within 2 months prior to randomization, requiring hospitalization for intravenous antibiotics or antiviral drug treatment;
* Live vaccine within 4 weeks prior to randomization or planned live vaccine during the study;
* Clinically significant infection, including but not limited to upper respiratory tract infection, lower respiratory tract infection, herpes simplex, herpes zoster, during the screening period, and requiring antibiotic or antiviral medication treatment;
* Has any significant illness or unstable clinical condition (such as renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurological, immune, or locally active infectious/infectious disease) that is judged by the investigator to be unsuitable for participation in this study.
* Abnormal laboratory tests during the screening period:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times upper limit of normal (ULN);
  2. Hemoglobin <90g/L;
  3. White blood cell count< 3.0×109/L;
  4. Neutrophil count<1.0×109/L;
  5. Lymphocyte count<0.5×109/L;
  6. Platelet count < 100×109/L;
  7. Total bilirubin >2 times ULN;
  8. Other significant laboratory test abnormalities that, in the opinion of the investigator, the subject is not suitable for participation in this study.
* History of malignant tumors (including carcinoma in situ) and lymphoproliferative disorders within 5 years prior to randomization;
* Those who have received at least 6 consecutive months of anti-IL-12, IL-17, IL23 monoclonal antibody drugs (such as ustekin, secukziu, ichizzo, gusechiu, etc.) at the approved dose but have poor clinical response (defined as not achieving PASI 50 during treatment)；
* Receipt of any other marketed or investigational biologic agent within 3 months or 5 half-lives (whichever is longer) prior to randomization;
* Receipt of any other investigational drug in 1 month or 5 half-lives (whichever is longer) prior to randomization;
* Those who have undergone surgical surgery within 4 weeks prior to randomization, or who plan to undergo surgical procedures during the study;
* Those who have lost blood or donated more than 400 mL of blood within 4 weeks prior to randomization;
* Receipt of immunoglobulin or blood products within 4 weeks prior to randomization;
* Systemic treatment drugs or immunosuppressants for psoriasis within 4 weeks prior to randomization, including but not limited to retinoids, glucocorticoids, methotrexate, cyclosporine, azathioprine, Janus kinase (JAK) inhibitors, etc;
* Use of strong CYP450 inducers (such as rifampicin, phenobarbital, carbamazepine, phenytoin, etc.) within 4 weeks prior to randomization;
* Received topical or systemic phototherapy within 4 weeks prior to randomization, including but not limited to Narrow-band ultraviolet B (NB-UVB), photochemotherapy (PUVA), 308nm excimer light;
* Use of topical drugs that may affect the severity of skin lesions in psoriasis within 2 weeks prior to randomization, including but not limited to glucocorticoids, urea, >3% salicylic acid, α or β hydroxy acids, retinoids, vitamin D3 analogues, calcineurin inhibitors, Phosphodiesterase-4 (PDE-4) inhibitors, etc. (Note: Mild emollients (without active substances such as urea, salicylic acid, α, or β hydroxy acids) are allowed to be used at all sites, but should not be used within 24 hours prior to each study visit);
* Potential difficulty in blood collection, with a history of fainting needle and blood sickness;
* Allergy to any of the known ingredients of the TQH3906, or any previous history of severe drug allergies.
* Those with a history of substance abuse;
* Has any other reasonable medical, psychiatric, or social reason that, in the opinion of the investigator, precludes participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving Psoriasis Area and Severity Index (PASI) 75 at week 12 | Up to week 12
  Achieve a PASI 75 ratio

SECONDARY OUTCOMES:
Proportion of patients achieving Static Physician's Global Assessment (sPGA) 0/1 at week 12 | Up to week 12
  It is used to observe the proportion of patients with 0 or 1
Proportion of patients achieving PASI 50 at week 12 | Up to week 12
  Observed proportion of patients achieving PASI 50 at week 12
Proportion of patients achieving PASI 90 at week 12 | Up to week 12
  Observed proportion of patients achieving PASI 90 at week 12
Proportion of patients achieving PASI 100 at week 12 | Up to week 12
  Observed proportion of patients achieving PASI 100 at week 12
Body Surface Area (BSA) score | Up to week 12
  To observe the degree of change from baseline in BSA score at week 12
Dermatology Life Quality Index (DLQI) score | Up to week 12
  To observe the degree of change from baseline in DLQI score at week 12
Incidence of abnormal laboratory test markers | From randomization to 4 weeks after the last dose
  The proportion of patients with abnormal laboratory examination indicators, including blood routine and liver function, mainly includes blood routine, liver function, etc.
Adverse event (AE) | From randomization to 4 weeks after the last dose
  Proportion of patients with adverse events, defined by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Serious Adverse Events (SAEs) | From randomization to 4 weeks after the last dose.
  Proportion of patients with serious adverse events, defined by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Tmax, ss | Within 1 hour before Day1, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day 15, Day 29, Day 57, Day 85 within 1 hour before administration, 1,1.5, 2, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours after Day 85
  Refers to the time when the blood concentration reaches its peak after a single dose. At this point in time, the blood concentration is the highest.
Cmax, ss | Within 1 hour before Day1, 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day15, Day29, Day57, Day85 within 1 hour before administration, and 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24, 48, 72 hours after Day85
  The steady-state concentration of the drug after multiple doses was investigated.
  Within 1 hour before Day1, 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day15, Day29, Day57, Day85 within 1 hour before administration, and 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24, 48, 72 hours after Day85.
Cmin, ss | Within 1 hour before Day1, 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day15, Day29, Day57, Day85 within 1 hour before administration, and 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours after Day85
  The lowest concentration from the initial moment after administration to the lowest concentration before the next dose when multiple doses reach steady state. This index is a common indicator to reflect the level of drug accumulation, and is closely related to the drug dose, dosing interval and drug elimination rate.
Area under the plasma concentration-time curve (AUC) 0-τ | Within 1 hour before Day1 administration, 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day15, Day29, Day57, Day85 within 1 hour before administration, and 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours after Day85
  When multiple administrations reach steady state, the area under the plasma concentration curve of each dosing interval is equal to the area under the plasma concentration curve from the time after administration to infinity.
Rac | Within 1 hour before Day1 administration, 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours, Day15, Day29, Day57, Day85 within 1 hour before administration, and 1 hour, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours after Day85
  The ratio of the dose required to be given in one dose to the total dose required to be given in divided doses.
Interleukin-17A (IL-17A) in serum | Within 1 hour before Day1 administration, Day15, Day29, Day85
  Change from baseline in serum IL-17A
Interleukin 19 (IL-19) in serum | Within 1 hour before Day1 administration, Day15, Day29, Day85
  Change from baseline in serum IL-19
β defensin in serum | Within 1 hour before Day1 administration, Day15, Day29, Day85
  Change from baseline in serum β defensin

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The first affiliated hospital of chongqing medical university, Chongqing, Chongqing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Liuzhou People'S Hospital, Liuchow, Guangxi
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital Of Xingtai Medical Colledge, Xingtai, Hebei
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang First People'S Hospital, Nanyang, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Wuhan First Hospital, Wuhan, Hubei
  - The First People's Hospital of Changde, Changde, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Hospital of Dermatology, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Genertec Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The first hospital of china medical university, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong First Medical University Affiliated Dermatology Hospital, Jinan, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Qingdao Municipal hospital (group), Qingdao, Shandong
  - Qingdao Traditional Chinese Medicine Hospital, Qingdao, Shandong
  - Shanghai JiaoTong University of medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - Affiliated Hangzhou First People'S Hospital,School of Medicine, Westlake University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang